CLINICAL TRIAL: NCT06698744
Title: A Phase 1 Single Arm, Open Label Study to Evaluate the Safety of UF-KURE-BCMA CAR-T Cells in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: UF-KURE-BCMA CAR-T Cells in Patients With Relapsed or Refractory Multiple Myeloma
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: David Wald (Other)
Responsible Party: Sponsor-Investigator, David Wald, Co-Leader, Immune Oncology Program, Case Comprehensive Cancer Center, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE1A24
Record Dates: First submitted 2024-11-07; First posted 2024-11-21 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Multiple Myeloma, Refractory
Keywords: UF- KURE-BCMA
MeSH Terms: conditions — Multiple Myeloma | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Intervention Model Description: Phase 1 single arm, open label study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- UF-KURE-BCMA T cell-based immunotherapy (Experimental): Pre-infusion will include multiple myeloma testing, preCAR-T evaluation, and cells will be collected. Participants will undergo lymphodepletion and inpatient CAR T-cell infusion. Patients will be monitored closely during a 28 day dose limiting toxicity (DLT) period.
  Interventions: Biological: UF-KURE-BCMA CAR T-cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: UF-KURE-BCMA CAR T-cells — Experimental anti-BCMA CAR T-cells manufactured with a proprietary ultrafast process. Patients will receive a single dose of CAR T-cells at one of three potential doses:
  * Dose -1: 3x10^6 cells
  * Dose 1: 10x10^6 cells
  * Dose 2: 15x10^6 cells
  Other Names: UF-KURE-BCMA cells
Drug: Cyclophosphamide — Patients will receive 3 days of intravenous (IV) cyclophosphamide 500 mg/m^2 days -5 to -3 or -4 to -2 where day 0 is the day of CAR T-cell infusion.
Drug: Fludarabine — Patients will receive 3 days of IV fludarabine 30 mg/m2 days -5 to -3 or -4 to -2 where day 0 is the day of CAR T-cell infusion.

SUMMARY:
The purpose of this study is to determine if UF-KURE-BCMA (B-Cell Maturation Antigen) chimeric antigen receptor T cells (CAR-T cells) can be used to treat relapsed or treatment refractory multiple myeloma (RRMM). This treatment uses T cells already present within the body that have been modified outside of the body by a virus and then returned by an infusion to fight cancer. The investigators are evaluating UF-KURE-BCMA because it uses a manufacturing process that is shorter than other Food and Drug Administration (FDA) approved CAR-T cells and only requires a simple blood draw. The standard treatments require weeks to manufacture the cells as well a special procedure to get an individual's cells. While the shorter manufacture time can be an advantage, the safety of this approach has not been demonstrated. The use of UF-KURE-BMCA is investigational and is not approved by the FDA outside of clinical trials. This is the first study of UF-KURE-BCMA in patients.

Participants will give a pint of blood, which is the amount one would provide if they were to donate blood. The blood will be used to make the UF-KURE-BCMA cells. Participants will then receive chemotherapy followed by a one-time infusion of the experimental modified CAR-T cells. After this infusion, participants will be watched for side effects and follow up will continue for up to 15 years.

DETAILED DESCRIPTION:
UF-KURE-BCMA is an autologous CAR-T cell therapy consisting of autologous cluster of differentiation 4 (CD4) positive and cluster of differentiation 8 (CD8) positive human T cells that are genetically engineered using a novel ultrafast lentiviral manufacturing system to express a humanized BCMA CAR-T that targets the BCMA receptor to eliminate multiple myeloma cells using simple peripheral blood draws instead of invasive leukapheresis. This ultrafast platform optimizes CAR-T potency and allows for quicker and cheaper manufacturing of these agents. The goal of this phase 1 study is to find recommended phase 2 dose of UF-KURE-BCMA for treatment of patients with relapsed or refractory multiple myeloma

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 years or older.
* Subjects must have Multiple Myeloma that is relapsed (defined as non-responsive or progressive disease while on therapy or within 60 days of last treatment in participants who had achieved a minimal response (MR) or better on prior therapy) after three or more lines of therapy including at least one proteasome inhibitor, one imide, and one anti-CD38 agent.
* Participants with multiple myeloma with comorbid amyloid and/or extramedullary disease will be eligible.
* To be eligible for response assessment, participants must have measurable disease at the time of screening defined as serum protein electrophoresis M-spike greater than or equal to 0.5 g/dl, urine protein electrophoresis M spike greater than or equal to 200 mg/24 hr, or difference in involved free light chain level of greater than or equal to 10 mg/dl provided serum free light chain (FLC) ratio is abnormal.
* ECOG Performance status ≤ 2
* Minimum of 2 weeks since prior radiation therapy or systemic therapy to treat malignancy at the time of blood sample collection for CAR-T manufacturing unless treatment was investigational, in which case a minimum of 4 weeks since last treatment is required. Prior CAR-T therapy is acceptable if participants exhibited progression free survival of greater than 6 months post CAR-T infusion.
* Total bilirubin ≤ 2X institutional upper limit of normal (except in participants with Gilbert's syndrome).
* AST (SGOT)/ALT (SGPT) ≤ 2.5 X institutional upper limit of normal.
* Calculated creatinine clearance ≥ 30mL/min estimated by the Cockcroft - Gault formula.
* Cardiac ejection fraction of ≥45% as determined by an echocardiogram.
* Adequate pulmonary function, defined as ≤ Grade 1 dyspnea and oxygen saturation (SaO2) ≥ 92% on room air. If pulmonary function tests (PFTs) are performed based on the clinical judgment of the treating physician, participants with forced expiratory volume in 1 second (FEV1) ≥ 50% of predicted and diffusing capacity for carbon monoxide (DLCO) (corrected for hemoglobin) of ≥ 40% of predicted will be eligible.
* Participants (or legal guardians) must have the ability to understand and the willingness to sign a written informed consent document.
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use a contraceptive method with a failure rate of < 1% per year during the treatment period and for at least 6 months after the UF-KUREBCMA CAR-T cell infusion. A woman is considered to be of childbearing potential if she is < 60 years old, postmenarcheal, has not reached a postmenopausal state (< 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus). Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below: With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after the UF-KURE-BCMA CAR-T cell infusion. Men must refrain from donating sperm during this same period. With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the UF-KURE-BCMA CAR-T cell infusion to avoid potential embryonal or fetal exposure. The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception.

Exclusion Criteria:

* Autologous stem cell transplant within 6 weeks of informed consent.
* Active CNS involvement of multiple myeloma.
* Plasma cell leukemia
* History of allogeneic hematopoietic stem cell transplantation.
* Second active malignancy, other than non-melanoma skin cancer or carcinoma in situ (e.g. cervix, bladder, breast). Stage 1 uterine cancer or localized prostate cancer.
* New York Heart Association class IV congestive heart failure.
* Cardiovascular disorders including unstable angina pectoris, clinically significant cardiac arrhythmias, myocardial infarction or stroke (including transient ischemic attack, or other ischemic event) within 6 months prior to registration.
* Known human immunodeficiency virus infection or acquired immunodeficiency syndrome related illness.
* Pregnant or breastfeeding women are excluded from this study because CAR-T cell therapy may be associated with the potential for teratogenic or abortifacient effects. Women of childbearing potential must have a negative serum pregnancy test. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with CAR-T cells, breastfeeding should be discontinued. These potential risks may also apply to other agents used in this study.
* Evidence of myelodysplasia or cytogenetic abnormality indicative of myelodysplasia on the most recent bone marrow biopsy prior to initiation of therapy.
* Serologic status reflecting active hepatitis B or C infection. Participants that are positive for hepatitis B core antibody, hepatitis B surface antigen (HBsAg), or hepatitis C antibody must have a negative polymerase chain reaction (PCR) prior to enrollment. (PCR positive participants will be excluded).
* Participants with history of clinically relevant CNS pathology such as epilepsy, seizure disorders, paresis, aphasia, uncontrolled cerebrovascular disease, severe brain injuries, dementia and Parkinson's disease.
* Participants with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, pulmonary abnormalities or psychiatric illness/social situations that would limit compliance with study requirements.
* History of active autoimmune disease (i.e. rheumatoid arthritis, systemic lupus erythematosus) with requirement of systemic immunosuppressive medications other than low dose steroids [i.e. maximum of 15mg prednisone equivalent] within the last 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12-11 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
To recommend a phase two cell dose for UF-KURE-BCMA. | 28 days
  Patients will be enrolled sequentially using a 3+3 design no sooner than every 28 days during the dose escalation phase and monitored for excessive dose limiting toxicities (DLT). If more than one DLT is observed in 6 patients treated, that dose is considered too toxic.
  The following serious adverse events are deemed DLTs. DLTs are graded per CTACAE V5 or ASTCT grading for CRS or ICANS.
  * Any death unless due to disease progression
  * Grade 4 CRS.
  * Grade 3 CRS that does not improve to ≤ grade 2 in 72 hours after treatment.
  * Grade 3 or higher ICANS.
  * Grade 4 neutropenia or thrombocytopenia that does not improve to ≤ Grade 2 within 42 days. Grade 3 thrombocytopenia with clinically significant bleeding.
  * Grade 3 or higher organ toxicity of any duration (Exception Grade 3 or 4 abnormal hepatic or renal function tests that improve to ≤ Grade 2 within 7 days).
  * All other Grade 3 toxicities, not attributable to disease or chemo that do not resolve to ≤ Grade 2 within 72 hours.
Incidence of trial stopping rule event | 28 days
  In the event of any of the following, study enrollment will be suspended pending safety review.
  1. Any treatment-related death (Grade 5 event) that occurs following treatment with UF-KURE-BCMA T cells and not related to disease progression.
  2. Unexpected severe toxicities such as
     1. Occurrence of Grade 4 DLTs in 2 subjects at the same dose level.
     2. Uncontrolled CAR T cell proliferation requiring CAR T cell ablation.
     3. Grade 4 neurotoxicity with cerebral edema.
     4. New malignancy distinct from recurrence/progression of previously treated malignancy and at least possibly related to IP.
     5. Replication-competent lentivirus (RCL) detection in any subjects.
  To re-initiate study enrollment, the sponsor and principal investigator will submit a study reactivation plan to the Food and Drug Administration for approval, including additional safeguards to prevent and minimize subsequent adverse events.

SECONDARY OUTCOMES:
Clinical responses of RRMM patients treated with UF-KURE-BCMA. | 90 days
  Clinical response will be defined by International Myeloma Working Group (IMWG) consensus response criteria using MM disease serologies, % bone marrow plasma cells, and next-generation sequencing MRD testing obtained at 30, 60, and 90 days post CAR-T infusion.
Median duration of response (DOR) in RRMM patients treated with UF-KURE-BCMA. | 2 years
  DOR will be defined as the time in months from the deepest clinical response as defined by IMWG criteria until disease progression or death, whichever comes first. Median DOR is the time at which 50% of patients have progressed.
Progression-free survival (PFS) in RRMM patients treated with UF-KURE-BCMA. | 2 year
  Progression free survival will be defined as the time from enrollment until either disease progression or death, which ever comes first. Median PFS will be defined as the time in months at which 50% of patients exhibit progressive disease or have died.
Feasibility of manufacturing UF-KURE-BCMA using peripheral blood. | 1 week
  Peripheral manufacturing of CAR T-cells from peripheral blood will be deemed feasible if the produced CAR T-product meets release criteria in 75% or more cases.
Overall survival (OS) in RRMM patients treated with UF-KURE-BCMA. | 2 years
  OS will be defined as the time from enrollment until death. Median OS will be defined as the time from enrollment in months at which 50% of patients have died.

CONTACTS AND LOCATIONS:
Overall Officials: James Ignatz-Hoover, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center Seidman Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Protocol, SAP and CSR will be shared.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Compiled and analyzed participant data will be published upon study completion. Publisher may request Protocol and Statistical Analysis Plan.
Access Criteria: Access criteria is not applicable